CLINICAL TRIAL: NCT02226146
Title: An Open-Label, Proof of Concept Study Designed to Evaluate the Safety, Efficacy and Pharmacodynamic Effect of Bertilimumab in Patients With Newly Diagnosed, Moderate to Extensive Bullous Pemphigoid
Brief Title: Evaluation of Safety, Efficacy and Pharmacodynamic Effect of Bertilimumab in Patients With Bullous Pemphigoid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Immune Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immune/BRT/BP-01
Record Dates: First submitted 2014-07-27; First posted 2014-08-27 (Estimated); Results first posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Pemphigoid, Bullous
Keywords: Pemphigoid Bullous; Bullous; Blisters; SKIN DISEASES; BP
MeSH Terms: conditions — Pemphigoid, Bullous; Blister; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bertilimumab (Experimental): Intravenous injection over 30 minutes of 10 mg/kg of Bertilimumab in physiological solution (PBS)
  Interventions: Biological: Bertilimumab

INTERVENTIONS:
Biological: Bertilimumab

SUMMARY:
This is an open-label, proof-of-concept, single group study in adult participants with newly diagnosed, moderate to extensive BP.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, ≥ 60 years of age.
2. Karnofsky performance status > 60%
3. Newly diagnosed, Bullous Pemphigoid per standard diagnostic criteria:

   * Clinical presentation [2]
   * Skin biopsy from a fresh blister showing subepidermal clefting and an inflammatory infiltrate consisting mainly of eosinophils
   * Immunofluorescence (IF) studies performed on uninvolved skin collected approximately 1 cm away from a fresh blister showing linear deposition of IgG and/or C3 along the basement membrane zone.
4. Moderate to extensive Bullous Pemphigoid defined by the mean number of new bullae and urticarial plaques that have appeared over the course of 3 days as determined by the investigator or referring physician (moderate disease defined by > 1 and ≤ 10 new bullae daily and ≥ 5 urticarial plaques and extensive disease by >10 new bullae daily) [3].
5. Adequate cardiac, renal and hepatic function as determined by the Investigator and demonstrated by screening laboratory evaluations, vital sign measurement, ECG recording and physical examination results.
6. Females of childbearing potential must agree to use effective contraception consistently throughout the study (such as hormonal contraception or two forms of barrier contraception) and have a negative serum pregnancy test at screening and a negative urine pregnancy test per the schedule of visits. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of amenorrhea or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks previously.
7. Males must have had a vasectomy or have expressed that they have no interest in fertility in the future.
8. Fertile males must agree to use effective contraception consistently throughout the study and for a period of four months following the end of study drug administration.
9. Willing and able to adhere to the study visit schedule and other protocol requirements.
10. Willing and able to provide voluntary written informed consent or written informed consent from a legally authorized representative with assent from the patient.

Exclusion criteria:

1. Patients with severe medical or surgical conditions at screening or baseline including, but not limited to, severe dementia or mental impairment, severe stroke, severe cardiac insufficiency, severe arterial hypertension, severe or uncontrolled renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, cerebral, psychiatric, or any other severe acute or chronic medical condition that may increase the risk associated with study participation/treatment or may interfere with the interpretation of study results and, in the Investigator's opinion, would make the patient inappropriate for study entry.
2. Presence of any malignancy that has been under active treatment (e.g., radiotherapy or chemotherapy) within the 2 years prior to baseline or is anticipated to require treatment during the study period (including follow up) with the exception of patients with removal of uncomplicated basal cell carcinoma or cutaneous squamous cell carcinoma, who may take part in the study.
3. Congenital or acquired immunodeficiency (e.g., common variable immunodeficiency, organ transplantation).
4. Clinically significant vital sign measurements or ECG findings as determined by the Investigator.
5. Clinically significant abnormal laboratory test results, unless regarded by the Investigator as related to BP, including but not limited to:

   * Hemoglobin level <10.0 g/dL
   * White blood cell count < 3 x 103/μL
   * Lymphocyte count < 0.5 x 103/μL
   * Platelet count <100 x 103/μL or >1200 x 103/μL
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 the upper limit of normal (ULN)
   * Alkaline phosphatase >3 ULN
   * Serum creatinine >2 ULN
6. Patients with mild, relapsed or refractory Bullous Pemphigoid. Mild disease defined by the mean number of new lesions that have appeared over the course of 3 days as determined by the investigator or referring physician, as follows: ≤ 1 bulla or < 5 urticarial plaques.
7. Concomitant skin conditions preventing physical evaluation of Bullous Pemphigoid.
8. Active or recent history of clinically significant infection within 1 month of baseline.
9. Pregnant or breast-feeding, or planning to become pregnant during the study.
10. Participation in a clinical trial of an investigational (unapproved) product within 4 weeks of baseline.
11. Known hypersensitivity to bertilimumab or any of the drug excipients.
12. Use of prednisone or other systemic steroids (excluding inhaled or ocular use of steroids) within 4 weeks prior to baseline. (Concomitant oral corticosteroids administered as part of the study protocol, from Day 0 onward, are allowed). Use of class 1 and 2 topical steroids (such as clobetasol propionate cream, reference Appendix D for further guidance) within 4 weeks prior to baseline. (Use of other topical steroids is allowed throughout the study at the discretion of the investigator).
13. Treatment with immunosuppressants (e.g., azathioprine, methotrexate) within 4 weeks prior to baseline.
14. Treatment with biologics (e.g., etanercept, adalimumab, ustekinumab, infliximab, intravenous Ig) within 4 months of baseline. Patients who have received rituximab within 1 year of baseline will be excluded from study participation.
15. Treatment with macrolides or tetracyclines within 4 weeks prior to baseline.
16. Received a vaccine or other immunostimulator within 4 weeks prior to baseline. Subject has current clinical, radiographic or laboratory evidence of active mycobacterium tuberculosis (TB) infection or prior evidence of active TB that, in the opinion of the investigator, has not been adequately treated or controlled and that represents a reactivation risk. If in the investigator's opinion the patient is at risk for latent TB, the patient should be evaluated for active/latent TB as applicable (e.g. PPD, QFT, and/or chest x-ray).

18. Evidence of an active disease of hepatitis B (HBsAg positive or HBcAb positive) or hepatitis C (HCV ab positive), CMV (IgM positive) or human immunodeficiency virus (HIV) infection (HIV1/2 Ab positive 19. Active abuse of alcohol or drugs. 20. Any other condition, which in the opinion of the Investigator would place the patient at an unacceptable risk if participating in the study protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (6):
  - Research Site, Iowa City, Iowa
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Salt Lake City, Utah
- Israel (2):
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Bertilimumab + Prednisone: Participants with moderate to extensive bullous pemphigoid (BP) received bertilimumab 10 milligrams/kilogram (mg/kg) intravenous (IV) infusion biweekly and prednisone at a maximum dose of 30 mg orally per the investigator's discretion.
Period: Overall Study
Arm/Group | Bertilimumab + Prednisone
Started | 11
Received at Least 1 Dose of Study Drug | 9
Completed | 8
Not Completed | 3
Not completed — Received rescue therapy | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The Safety analysis population consisted of all participants enrolled in the trial who received at least one infusion of bertilimumab 10 mg/kg.
Groups:
- Bertilimumab + Prednisone: Participants with moderate to extensive BP received bertilimumab 10 mg/kg IV infusion biweekly and prednisone at a maximum dose of 30 mg orally per the investigator's discretion.
Arm/Group | Bertilimumab + Prednisone
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity has not been collected.
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 8
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Anti-Drug Antibodies
Time Frame: Baseline up to 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Bertilimumab + Prednisone
Number analyzed (Participants) | 9
Participants | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant, which does not necessarily have a causal relationship with the study treatment. TEAEs were defined as AEs that started on or after the first administration of study drug until the end of the follow up period. A summary of serious and non-serious AEs regardless of causality is located in 'Reported Adverse Events module'.
Time Frame: Baseline up to 1 year
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Bertilimumab + Prednisone
Number analyzed (Participants) | 9
Participants | 6

3. Secondary Outcome: Number of Participants Who Achieved at Least 50%, 70% and 90% Reduction From Baseline in Total Activity Score of the Bullous Pemphigoid Disease Area Index (BPDAI) Score
Description: BPDAI is a clinician completed tool that is used for independent disease severity assessment to measure disease extent in bullous pemphigoid. The total BPDAI activity score was calculated as the arithmetic sum of the 3 subcomponents - cutaneous blisters/erosions, cutaneous urticaria/erythema, and mucosal blisters/erosions. The BPDAI total activity gives an indication of disease activity, with score range from 0 (no disease activity) to 360 (severe disease activity). Higher scores indicated greater disease activity. Baseline was defined as the last measurement obtained before the treatment initiation.
Time Frame: Baseline, Day 84
Population: The Efficacy population included all participants in the safety population who had the visit score on the BPDAI at baseline and at least one post baseline BPDAI score. Here, overall number of participants analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Bertilimumab + Prednisone
Number analyzed (Participants) | 7
Participants
  50% Reduction | 6
  70% Reduction | 5
  90% Reduction | 4

4. Secondary Outcome: Number of Participants Who Had Tapered to Prednisone Dose of ≤ 10 mg/Day
Time Frame: Baseline, Day 84
Population: The Efficacy population included all participants in the safety population who had the visit score on the BPDAI at baseline and at least one post baseline BPDAI score.
Measure: Count of Participants; unit: Participants
Arm/Group | Bertilimumab + Prednisone
Number analyzed (Participants) | 9
Participants | 5

5. Secondary Outcome: Percentage of Reduction From Baseline in BPDAI Pruritis (Visual Analogue Scale [VAS]) Total Score
Description: The VAS sub-scores were defined as: 1. VAS Sub-Score I: How severe has your itching been over the last 24 hours. 2. VAS Sub-Score II: How severe has your itching been over the past week. 3. VAS Sub-Score III: How severe has your itching been over the past month. The Total Pruritus VAS score was defined as the sum over the three sub-scores. If at least one of the sub-scores is missing, the total is not defined. If value for the pruritus total score could not be determined than the value was left as blank for the calculation of the mean. Scores for the BPDAI-VAS ranged from 0 to 30, with higher scores indicating a worse condition.
Time Frame: Baseline, Day 84
Population: as for outcome 4
Measure: Mean (Full Range); unit: percentage of reduction in BPDAI VAS
Arm/Group | Bertilimumab + Prednisone
Number analyzed (Participants) | 9
percentage of reduction in BPDAI VAS | 8.6 [3 to 19]

6. Secondary Outcome: Percentage of Reduction From Baseline in Autoimmune Bullous Diseases Quality of Life (ABQOL) Total Score
Description: ABQoL questionnaire assessed the impact of autoimmune bullous disease and their therapies on the daily life of participants. Scores range from 0 to 51 with a higher score representing a worse quality of life. If value for the ABQOL total score could not be determined than the value was left as blank for the calculation of the mean.
Time Frame: Baseline, Day 84
Population: as for outcome 4
Measure: Mean (Full Range); unit: percentage of reduction in ABQOL score
Arm/Group | Bertilimumab + Prednisone
Number analyzed (Participants) | 9
percentage of reduction in ABQOL score | 11 [1 to 39]

ADVERSE EVENTS:
Time Frame: Baseline up to 1 year
Description: The Safety analysis population consisted of all participants enrolled in the trial who received at least one infusion of bertilimumab 10 mg/kg.
Arm/Group | Bertilimumab + Prednisone
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bertilimumab + Prednisone (N=9)
Peripheral vascular disorder (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bertilimumab + Prednisone (N=9)
Blurred vision (Eye disorders) | 1
Traumatic laceration right big toe (Injury, poisoning and procedural complications) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Night sweating (Reproductive system and breast disorders) | 1
Edema (bilateral) (General disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gamma-Glutamyl Transferase increased (Hepatobiliary disorders) | 1
Cyst at base of tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

LIMITATIONS AND CAVEATS:
Study conducted by Immune Pharmaceuticals Inc. and was acquired by Alexion Pharmaceuticals, Inc after study completion, database lock, and report generation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-02-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT02226146/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/46/NCT02226146/SAP_001.pdf